CLINICAL TRIAL: NCT03743181
Title: Impact of Clinical Pharmacy Services Provided for Patients With Active Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: hager omar mohammed siddik (Other)
Responsible Party: Sponsor-Investigator, hager omar mohammed siddik, Teaching assistant at clinical pharmacy department at faculty of pharmacy ain shams university, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: 156
Record Dates: First submitted 2018-11-04; First posted 2018-11-16 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Pharmaceutical Services

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- intervention: will be supplied by pharmaceutical care services provided by the clinical pharmacist plus standard care by physician in attendance.
  Interventions: Other: pharmaceutical care services
- control: will received standard care by physician in attendance

INTERVENTIONS:
Other: pharmaceutical care services — detection of drug therapy problems and investigation of the impact of clinical pharmacist interventions on the patient clinical outcome and quality of life
  Groups: intervention

SUMMARY:
Enrolment of clinical pharmacy services in RA patients as a part of health care system has been investigated at many studies but not investigated in active RA patients before. This study aimed to detect drug therapy-related problems (DTRPs) in active rheumatoid arthritis (RA) patients and Investigate the impact of clinical pharmacist interventions on the patient clinical outcome and quality of life (QoL). Methods:Prospective, randomized controlled study to be carried out at rheumatology outpatient clinic, Ain Shams University Hospitals on 50 patients with active RA for 6 months.determine if any drug therapy problems are present.Develop a plan of care that includes interventions to resolve drug therapy problems, achieve goals of therapy, and prevent drug therapy problems. questionnaires was used to measure functional status in RA patients using health assessment questionnaire (HAQ) and assess self-reported quality of life in patients with (RA) using rheumatoid arthritis quality of life questionnaire (RAQOL) and measure adherence using the 4-item Morisky Green Levine Medication Adherence Scale and Disease Activity Score-28 was used as an objective method to assess RA disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-60 years old
* fulfillment of the American College of Rheumatology /European league against rheumatism (2010 ACR/EULAR ) diagnostic criteria for RA.
* patients with active RA(defined by DAS28 score < 5.1)

Exclusion Criteria:

* Patients with cognitive impairment.
* The presence of hepatic or renal disease.
* The presence of other rheumatic and connective tissue disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: rheumatoid arthritis patients from outpatient clinics - Ain shams university hospitals
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2018-01-14 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
disease activity score | 6 months
  disease activity score-28 (DAS-28) for measuring disease activity in rheumatoid arthritis patients
Quality of life questionnaire | 6 months
  Rheumatoid arthritis quality of life questionnaire (RAQOL) for measuring quality of life
Health assessment questionnaire | 6 months
  Health assessment questionnaire (HAQ) for measuring functional status in rheumatoid arthritis patients

CONTACTS AND LOCATIONS:
Overall Officials: hager omar m siddik, Principal Investigator — teaching assistant at faculty of pharmacy ain shams university
Locations (1):
- Facuty of Pharmacu Ain Shams University, Cairo, Abasiya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided